CLINICAL TRIAL: NCT00760838
Title: The AZIthromycin in Severe ASThma (AZISAST) Study: a Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study Evaluating the Efficacy, Safety and Cost-effectiveness of Azithromycin as add-on Therapy in Adult Subjects With Severe Persistent Asthma, Who Remain Inadequately Controlled Despite GINA (2006) Step 4 or 5 Therapy
Brief Title: AZISAST Study: AZIthromycin in Severe ASThma Study
Acronym: AZISAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008/445; IWT 070709
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Asthma
Keywords: Inadequately controlled severe asthma
MeSH Terms: conditions — Asthma | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azithromycin (Experimental): Azithromycin 250 mg
  1x/day during 5 days 3x/week afterwards
  Interventions: Drug: Azithromycin 250 mg
- placebo (Placebo Comparator): Placebo
  1x/day during 5 days 3x/week afterwards
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin 250 mg — Azithromycin 250 mg three times a week during treatment period (6 months); run-in period of 2 weeks; wash-out period of 4 weeks
  Arms: Azithromycin
Drug: Placebo — Placebo three times a week during treatment period (6 months); run-in period of 2 weeks; wash-out period of 4 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and cost-effectiveness of azithromycin as add-on therapy in adult subjects with severe persistent asthma, who remain inadequately controlled despite GINA (2006) step 4 or 5 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. patients who have given written informed consent
2. males or females of any race
3. 18-75 years of age
4. with the diagnosis of persistent asthma ≥ 1 year duration at screening and a history consistent with GINA step 4 or 5 clinical features
5. receiving high dose ICS plus inhaled LABA for at least 6 months prior to screening
6. patients who have suffered multiple (i.e. at least two) independent documented severe asthma exacerbations within the previous 12 months
7. patients must be never-smokers or ex-smokers with a smoking history of ≤ 10 pack-years.

Exclusion Criteria:

1. females who are pregnant or who are breastfeeding
2. patients with severe bronchiectasis
3. patients with active tuberculosis or non-tuberculous mycobacterial infections (NTM)
4. patients with significant underlying medical conditions (e.g. infection, hematological disease, malignancy, neurologic, renal, hepatic, coronary heart disease or other cardiovascular disease, endocrinologic or gastrointestinal disease) within the previous 3 months
5. who are unable to perform spirometry or complete a patient diary or complete questionnaires
6. patients with known hypersensitivity to azithromycin or other macrolide antibiotics
7. patients who's heart rate corrected QT interval is prolonged
8. patients who have - in the judgement of the investigator - a clinically relevant laboratory abnormality
9. patients currently treated with macrolide antibiotics or recent macrolide treatment (in the past twelve weeks)
10. anti-IgE treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Brusselle, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (7):
- Belgium (7):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - ZNA Middelheim, Antwerp
  - AZ Sint-Jan Brugge, Bruges
  - Ghent University Hospital, Ghent
  - AZ Groeninge, Kortrijk
  - Universitair Ziekenhuis Leuven, Leuven
  - AZ Heilig Hart Roeselare, Roeselare

REFERENCES:
- [Derived] Undela K, Goldsmith L, Kew KM, Ferrara G. Macrolides versus placebo for chronic asthma. Cochrane Database Syst Rev. 2021 Nov 22;11(11):CD002997. doi: 10.1002/14651858.CD002997.pub5. PMID 34807989
- [Derived] Brusselle GG, Vanderstichele C, Jordens P, Deman R, Slabbynck H, Ringoet V, Verleden G, Demedts IK, Verhamme K, Delporte A, Demeyere B, Claeys G, Boelens J, Padalko E, Verschakelen J, Van Maele G, Deschepper E, Joos GF. Azithromycin for prevention of exacerbations in severe asthma (AZISAST): a multicentre randomised double-blind placebo-controlled trial. Thorax. 2013 Apr;68(4):322-9. doi: 10.1136/thoraxjnl-2012-202698. Epub 2013 Jan 3. PMID 23291349
- See also: Website of the Ghent University Hospital — http://www.uzgent.be

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Azithromycin
Started | 54 | 55
Completed | 49 | 53
Not Completed | 5 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Azithromycin | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 55 | 109
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [36 to 60] | 53 [46 to 64] | 53 [46 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 29 | 67
  Male | 16 | 26 | 42
Region of Enrollment [Number; unit: participants]
  Belgium | 54 | 55 | 109

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Severe Asthma Exacerbations
Description: Severe asthma exacerbations are defined as severe asthma episodes for which a treatment with antibiotics or cortisone is administered for a minimum of 3 days.
Time Frame: from baseline to week 26
Population: intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 54 | 55
proportion of participants | 0.52 [0.36 to 0.75] | 0.55 [0.38 to 0.78]

2. Secondary Outcome: Proportion of Participants Using Rescue Medication From Baseline to Week 26
Description: proportion of participants using rescue medication is defined as the the number of participants who had to use rescue medication from baseline untill week 26, independent on the number of times the medication had to be used.
  This measure was conducted by averaging the proportion of participants using rescue medication from each week between baseline and week 26.
Time Frame: from baseline to week 26
Population: intention to treat analysis
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 54 | 55
proportion of participants | 0.24 (2.11) | 0.08 (1.14)

3. Secondary Outcome: Peakflow Measurements
Description: change in peak expiratory volume peak expiratory volume is measured as a maximal expiration for 1 second
Time Frame: from baseline to week 26
Population: intention to treat analysis
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 54 | 55
L/min
  morning Peak Expiratory Volume | -5.77 (48.20) | -1.81 (54.27)
  evening Peak Expiratory Volume | -4.65 (78.68) | -0.81 (48.47)

4. Secondary Outcome: Change in Forced Expiratory Volume in 1 Second
Time Frame: from baseline to week 26
Population: intention to treat analysis
Measure: Mean (Standard Deviation); unit: percentage of baseline FEV1
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 54 | 55
percentage of baseline FEV1
  pre-bronchodilatator FEV1 | -0.90 (11.79) | -0.02 (10.06)
  post-bronchodilatator FEV1 | -0.66 (1.29) | 8.84 (12.50)

5. Secondary Outcome: Change in Total Score on Asthma Control Questionnaire (ACQ)
Description: A simple questionnaire to measure the adequacy of asthma control and change in asthma control which occurs either spontaneously or as a result of treatment.
  ACQ has a multidimensional construct assessing symptoms (5 items--self-administred) and rescue inbronchodilator use (1 item-self-administered), and FEV1% (1 item) completed by clinic staff
  Scaling of items: 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 categories for FEV1%)
  Scores range between 0 (totally controlled) and 6 (severely uncontrolled).
Time Frame: from baseline to week 26
Population: intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 54 | 55
units on a scale | -0.12 (0.70) | -0.24 (0.93)

6. Secondary Outcome: Change in Total Score on the Asthma-related Quality of Life (AQLQ)
Description: A disease-specific health-related quality of life instrument that taps both physical and emotional impact of disease
  32 items with 2-week recall: Symptoms (11 items), Activity Limitation (12 items, 5 of which are individualized), Emotional Function (5 items), and Environmental Exposure (4 items)
  7-point Likert scale (7 = not impaired at all - 1 = severely impaired).
  Scores range 1-7, with higher scores indicating better quality of life.
Time Frame: from baseline to week 26
Population: intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 54 | 55
units on a scale | 0.20 (0.73) | 0.32 (0.89)

ADVERSE EVENTS:
Time Frame: from randomisation to exit visit (during the whole study period, at least 24 weeks)
Arm/Group | Placebo | Azithromycin
Serious Adverse Events (participants affected / at risk) | 4/54 | 7/55
Other Adverse Events (participants affected / at risk) | 39/54 | 37/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Azithromycin (N=55)
deep venous trombosis (Blood and lymphatic system disorders) | 0 (0) | 1
cerebrovascular accident (Blood and lymphatic system disorders) | 0 | 1
gastro-enteritis (Gastrointestinal disorders) | 0 | 1
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 | 3
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
acute myocardial infarction (Cardiac disorders) | 1 | 0
oesophagitis grade A (Gastrointestinal disorders) | 0 | 1
pseudoparalysis right shoulder (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Azithromycin (N=55)
lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 22 (34) | 17 (24)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 27 (41) | 26 (40)
nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
headache (Nervous system disorders) | 3 (3) | 3 (4)
diarrhea (Gastrointestinal disorders) | 7 (8) | 3 (3)
abdominal pain (Gastrointestinal disorders) | 6 (8) | 2 (2)
vertigo (Nervous system disorders) | 1 (1) | 2 (2)
allergic reaction (Immune system disorders) | 1 (1) | 2 (2)
elevated liver function event (Hepatobiliary disorders) | 0 | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 (1)
leucopenia (Blood and lymphatic system disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes